CLINICAL TRIAL: NCT05824910
Title: Effect of Pulmonary Telerehabilitation and Telemonitoring for Patients With Chronic Respiratory Diseases: a Feasibility Study
Brief Title: Effect of Pulmonary Telerehabilitation and Telemonitoring for Patients With Chronic Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Principal Investigator, Diana C Sanchez-Ramirez, PhD, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25892 (B2023:030)
Record Dates: First submitted 2023-03-13; First posted 2023-04-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: COPD; Interstitial Lung Disease
Keywords: chronic respiratory diseases; telemonitoring; telerehabilitation; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: one group pre/post assessment (feasability study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Small group zoom meeting (Experimental): 2 groups of 6 participants will be asked to follow the exercise program with their peers in a zoom meeting 3 times a week for 45 min each time. This time includes 5 min before and 10 min after for free talk and chat between participants. There will also be a weekly zoom education session for 30min.
  Interventions: Other: Exercise program (virtual/remote)

INTERVENTIONS:
Other: Exercise program (virtual/remote) — Intervention (8 weeks): using the participants' initial assessment and personal characteristics, the therapist will provide personalized recommendations (e.g. maximum heart rate, minimum SpO2), explain the educational materials, and instruct patients on safety precautions

SUMMARY:
This research study is being conducted to evaluate the feasibility of using technology to deliver a remote home exercise program and assess the health outcomes of patients with chronic lung diseases. Specific objectives are to assess the interventions on patients: 1) Lung function, 2) Dyspnea, 3) Fatigue, 4) Exercise capacity, 5) Self-efficacy, and 6) Health-related quality of life. The investigators will also be evaluating the practicality of using videoconferencing and commercial wearable telemonitoring devices (ie. smart watches) for the implementation of the intervention in this group of patients.

DETAILED DESCRIPTION:
This feasibility study uses a one group pre-post intervention study. In a subsequent stage, the possibility of conducting a matched (age, gender, diagnosis) case-control study comparing the effects of this study with the current Pulmonary Rehab WRHA program on patients' outcomes will be explored.

Participants who meet the inclusion criteria will be invited to an initial assessment session of approximately 1 hour (week 0) at the RespirabilityLab (Riverview Health Centre - 4th floor of the Princess Elizabeth Building). A registered therapist in charge of implementing the intervention will request informed consent to participate in the study, explain specifics of the intervention to each participant, and will conduct an initial assessment. Using the participants' initial assessment and personal characteristics, the therapists will provide personalized recommendations (e.g. maximum heart rate, minimum SpO2), and instruct patients on safety precautions (how to pace themselves, when to seek professional or emergency care).

All will receive training in 1) basic device management (join a Zoom meeting, and apps needed), 2) use of a portable spirometer, pulse oximeter and smartwatch, and their associated apps.

Two groups of 6 patients will complete an 8-week program (2 rounds of 12 participants for a total of 24 participants in total). The exercise program will involve a small group of peers (2 groups/6 participants each) in a Zoom meeting 2 times a week/45 min each (including 5 min before and 10 min after the meeting for free talk-chat between the participants e.g. questions, perceptions, etc.). The RA will organize the Zoom meetings, will resolve general questions (e.g. equipment, platforms, etc.) and will act as a direct point of contact between the therapist and the participants. An education session (~30-45 min) will be offered to all participants (12 at a given time) once a week over the 8 weeks on key topics such as managing smoking cessation, managing shortness of breath, exercising with chronic lung disease, managing fatigue, etc. Patients will be asked to always wear a smartwatch and a pulse oximeter while exercising so that they can control their pace while avoiding exceeding target values (HR, Sp02). After each exercise session, participants will be asked to open apps on their smartphone or tablet linked to the wearable devices via Bluetooth so that the data can be transmitted to the research team (Labfront dashboard) or emailed to the RA (CVS format). Participants will be able to contact the therapist or the RA at any time during the study if they have questions or concerns. Otherwise, the patients will be contacted if abnormal values are identified in the telemonitoring data.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of COPD or ILD
* living in Manitoba
* Access to smart phone or tablet and home internet service

Exclusion Criteria:

* acute exacerbation of their condition
* history of neurological disease or mental illness
* inability to ambulate independently without supervision
* inability to complete basic tasks on a smart phone or tablet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Lung Function | 8 weeks
  % predicted FEV1 and FVC will be assessed using a SpiroBank Smart F/V multi parameter spirometer (MIR) at pre-post intervention and once a week in between to monitor changes. This portable spirometer, which is MDSAP approved and complaint with ATS/ ERS guidelines, connects automatically via Bluetooth to an iOS & Android compatible App (MIR Spirobank).
Change in Dyspnea | 8 weeks
  Modified Borg Scale (0 "best" to 10 "worse") will be used to assess dyspnea.
Change in Fatigue | 8 weeks
  Fatigue severity scale (0 -7 "higher worse") will be used to measure the severity of fatigue.
Change in Exercise Capacity | 8 weeks
  Assessed with the one-minute sit-to-stand test (number of times the persons can complete the task in one minute).
Change in Self-efficacy | 8 weeks
  Assessed using the Self-Efficacy for Managing Chronic Disease 6-Item Scale each rated from 0 "not at all confident" to 10 "totally confident")
Change in Health Relate quality of life | 8 weeks
  Assessed with the Clinical COPD Questionnaire (Scored from 0 - 6 [worse])
Change in Dyspnea severity | 8 weeks
  Assessed with the modified Medical Research Council (0-4 "higher is worse outcome").
Impact of cough on quality of life | 8 weeks
  Assessed with the Leicester Cough Questionnaire (3 - 21 points). Lower scores indicate higher impact of cough on quality of life
Level of Dysphagia | 8 weeks
  Assessed with the Sydney Swallow Questionnaire(0-100mm "higher represent worse outcome").
Change in Health Relate quality of life | 8 weeks
  Assessed with the St. George's Respiratory Questionnaire. Total score is calculated from 0 (no health impairment) to 100 (maximum health impairment)

SECONDARY OUTCOMES:
Participant feedback questionnaire | 8 weeks
  A questionnaire will be used to capture the participants' level of satisfaction with the study using a 5-points liker scale.

CONTACTS AND LOCATIONS:
Overall Officials: Diana C Sanchez-Ramirez, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada